CLINICAL TRIAL: NCT05953649
Title: Effect of Early Extracorporeal Diaphragm Pacing （EDP） Combined With Tilt Table Verticalization （TTV) on Diaphragm Function in Critically Ill Patients With Mechanical Ventilation: a Randomized Controlled Trial.
Brief Title: Effect of Early Extracorporeal Diaphragm Pacing Combined With Tilt Table in Ventilated Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2023-376-02
Record Dates: First submitted 2023-06-12; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-05

CONDITIONS: Early Mobilization; Critically Ill; Mechanical Ventilation; Diaphragm Dysfunction
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): In the control condition, patients received conventional physiotherapy (CPT) according to standard clinic procedures.
  Interventions: Other: Conventional Physiotherapy
- experimental group 1 (Experimental): the experimental group uses Extracorporeal Diaphragm Pacing (EDP) on the basis of the control group.
  Interventions: Device: Extracorporeal Diaphragm Pacing; Other: Conventional Physiotherapy
- experimental group 2 (Experimental): the experimental group used Extracorporeal Diaphragm Pacing (EDP) combined with Tilt Table Verticalization (TTV) on the basis of the control group.
  Interventions: Device: Extracorporeal Diaphragm Pacing; Device: Tilt Table Verticalization; Other: Conventional Physiotherapy

INTERVENTIONS:
Device: Extracorporeal Diaphragm Pacing — In the EDP group, a pacer using the extracorporeal diaphragm pacemaker provided by Guangzhou Xueliang Biotechnology Developing Co., Ltd., the pacing electrode is pasted on the body surface closest to the phrenic nerve at the outer edge of the lower end of the sternocleidomastoid muscle under ultrasound guidance, and the auxiliary electrode is placed between the second intercostal of the midline of the clavicle. The intensity of treatment parameters was set from low to high, and the intensity of treatment was increased when the patient could tolerate it, pacing 12-18 times/min at a frequency of 40 hertz (Hz)/30min/time, and performed every 12 hours for a week.
  Other Names: External Diaphragm Pacing
  Arms: experimental group 1; experimental group 2
Device: Tilt Table Verticalization — VitalGo bed (VitalGo Systems Ltd., Fort Lauderdale） is used for verticalization. Verticalization was set to minimum 30°, depending on cardiopulmonary parameters (respiratory rate, heart rate, blood pressure, oxygen saturation), vertical position was gradually increased (in 5° steps) to a maximum of 90°, as long as the above-named cardiopulmonary parameters of the patient remained stable and remain this position for 30 minutes simultaneously with extracorporeal diaphragm pacing for a week.
  Other Names: Tilt Table Standing; head-up tilt
  Arms: experimental group 2
Other: Conventional Physiotherapy — Patients receive early mobilization, which refers to a series of clinical intervention protocols (such as passive movement or active exercises, etc.) that confers physical benefits at an early period in collaboration with a multidisciplinary team (intensive care physicians, rehabilitation physicians, physical therapists, occupational therapists, respiratory therapists, and nurses). The study intervention take place during working time between 8 a.m. and 17 p.m. Patients of all three study groups receive this rehabilitation program until they transfer out of ICU.

SUMMARY:
The aim of this study is to test the effect of 1week of extracorporeal diaphragm pacing (EDP) combined either with or without tilt table verticalization (TTV) on diaphragm function in patients with mechanical ventilation compared to conventional physiotherapy (CPT).

DETAILED DESCRIPTION:
In order to explore whether extracorporeal diaphragm pacing (EDP) combined with tilt table verticalization (TTV) improves diaphragm function in mechanically ventilated patients, the investigators conducted a three-arms randomized controlled trial of 90 ventilated patients in the ICU of a general hospital in the southern China state of Guangzhou. After assessment of inclusion and exclusion criteria, patients were randomly assigned to one of the following three groups: (1) EDP with TTV and with conventional physiotherapy (CPT) (n = 30), (2) EDP without TTV and with CPT (n = 30), and (3) conventional physiotherapy (CPT; n = 30).

ELIGIBILITY:
Inclusion Criteria:

* Duration of mechanical ventilation prior to enrollment≤ 72 hours.
* Expected duration of mechanical ventilation≥72 hours.
* Participants (or their legal representatives) have signed informed consent.

Exclusion Criteria:

* Pregnancy or breast-feeding.
* Prone ventilation or current extracorporeal membrane oxygenation.
* Hemodynamic instability: mean arterial pressure is less than 65 millimeters of mercury (mmHg) or higher than 85 millimeters of mercury (mmHg), heart rate > 150 beats / minute, intravenous use of larger doses of vasopressors (such as dopamine > 10 mg/ (kg· min) or norepinephrine/epinephrine >0.1 mg/ (kg· min)) or aortic balloon counter pulsation; respiratory rate< 5 breaths per minute; Oxygen saturation< 88%.
* New-onset myocardial ischemia.
* Unstable cervical spine fracture and spinal cord injury.
* Deterioration of neurological function, requiring intracranial pressure monitoring and ventricular drainage, or active control of intracranial hypertension.
* Current neuromuscular block treatment or pre-existing neuromuscular disease or neuromuscular junction disease affecting respiratory muscle (such as myasthenia gravis, Guillain-Barré syndrome, etc.).
* There are contraindications to diaphragmatic pacing (local skin, tissue incompleteness or infection, chest X-ray examination shows pneumothorax or pleural effusion accounting for 1/3 of bilateral chest cavity).
* Body mass index (BMI) ⩾40 kg/m2.
* Known / suspected phrenic nerve palsy.
* Patients who refuse active treatment or are in the terminal stage of malignant tumors, have an expected life expectancy of < 6 months, etc.
* Participated in other clinical studies related to mechanical ventilation within 2 months prior to the start of the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-05-27 (Estimated); Study Completion 2024-07-27 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline on Diaphragm Thickening Fraction at Day 4 and Day 7. | Baseline, Day 4 and Day 7.
  The Diaphragm thickening fraction-DTf (%) was calculated as the difference between end-expiration and end-inspiration divided by end-inspiration × 100.Diaphragm thickening fraction (DTf) less than 20% is a measure of ultrasonographic diaphragmatic dysfunction in patients on mechanical ventilation.

SECONDARY OUTCOMES:
Change from Baseline on Ventilation mode at Day 4 and Day 7. | Baseline, Day 4 and Day 7.
  A ventilator mode is a way of describing how the mechanical ventilator assists the patient with taking a breath.
Change from Baseline on Positive End-expiratory Pressure (PEEP) at Day 4 and Day 7. | Baseline, Day 4 and Day 7.
  Positive end-expiratory pressure (PEEP) is the positive pressure that will remain in the airways at the end of the respiratory cycle (end of exhalation) that is greater than the atmospheric pressure in mechanically ventilated patients.
Change from Baseline on minute ventilation at Day 4 and Day 7. | Baseline, Day 4 and Day 7.
  It usually refers to the expired amount and can be calculated using the following equation: minute ventilation (VE)= tidal volume (VT) ×respiratory frequency(f)
Change from Baseline on tidal volume at Day 4 and Day 7. | Baseline, Day 4 and Day 7.
  Tidal volume is the amount of air that moves in or out of the lungs with each respiratory cycle.
Change from Baseline on Maximum Inspiratory Pressure (MIP） at Day 4 and Day 7. | Baseline, Day 4 and Day 7.
  The maximum inspiratory pressures measure the maximal efforts of the respiratory muscles.
Change from Baseline on airway occlusion pressure (P0.1) at Day 4 and Day 7. | Baseline, Day 4 and Day 7.
  P0.1 is a parameter for the neuro-muscular activation of the respiratory system, which is an important determinant for the work of breathing.
Change from Baseline on transdiaphragmatic pressure at Day 4 and Day 7. | Baseline, Day 4 and Day 7.
  Transdiaphragmatic pressure (Pdi) represents the pressure across the diaphragm, which can be expressed as the difference between abdominal pressure (Pab) and pleural pressure (Ppl):Pdi = Ppl- Pab.
Change from Baseline on MRC score at Day 4 and Day 7. | Baseline, Day 4 and Day 7.
  Medical Research Council (MRC)-sum score evaluates global muscle strength. Manual strength of six muscle groups (shoulder abduction, elbow flexion, wrist extension, hip flexion, knee extension, and ankle dorsiflexion) is evaluated on both sides using MRC scale. Summation of scores gives MRC-sum score, ranging from 0 to 60.
Change from Baseline on Blood oxygen status at Day 4 and Day 7. | Baseline, Day 4 and Day 7.
  Oxygenation Index = (FiO2× Mean Airway Pressure) / partial pressure of oxygen in arterial blood (PaO2) The oxygenation index is used to assess the intensity of ventilatory support required to maintain oxygenation.

OTHER OUTCOMES:
Day 28 mortality | within 28 days of the finishing of the trial.
  Short-term mortality was defined as a date of all-cause death within 28 days of the finishing of the trial.
ventilator free days | within 28 days of the start of the trial
  It is defined as a date of no ventilation within 28 days of the start of the trial.
Length of stay in ICU | up to 28 days.
  The patient's length of stay in the ICU since the beginning of inclusion.
Ratio of short weaning | within 28 days of the start of the trial
  It is defined as the first separation attempt resulted in a termination of the weaning process within 24 hours (successful separation or early death).
Duration of control ventilation | within 28 days of the start of the trial
  It is defined as the ventilation mode in which the frequency, tidal volume, and inspiratory time of breathing are controlled by a ventilator because the patient has no spontaneous breathing or very weak spontaneous breathing.
Duration of ventilation | within 28 days of the start of the trial
  It is defined as a date of ventilation within 28 days of the start of the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Zhijie He, Study Director — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University

REFERENCES:
- [Background] Berger D, Bloechlinger S, von Haehling S, Doehner W, Takala J, Z'Graggen WJ, Schefold JC. Dysfunction of respiratory muscles in critically ill patients on the intensive care unit. J Cachexia Sarcopenia Muscle. 2016 Sep;7(4):403-12. doi: 10.1002/jcsm.12108. Epub 2016 Mar 9. PMID 27030815
- [Background] Powers SK, Kavazis AN, Levine S. Prolonged mechanical ventilation alters diaphragmatic structure and function. Crit Care Med. 2009 Oct;37(10 Suppl):S347-53. doi: 10.1097/CCM.0b013e3181b6e760. PMID 20046120
- [Background] Levine S, Nguyen T, Taylor N, Friscia ME, Budak MT, Rothenberg P, Zhu J, Sachdeva R, Sonnad S, Kaiser LR, Rubinstein NA, Powers SK, Shrager JB. Rapid disuse atrophy of diaphragm fibers in mechanically ventilated humans. N Engl J Med. 2008 Mar 27;358(13):1327-35. doi: 10.1056/NEJMoa070447. PMID 18367735
- [Background] Supinski GS, Callahan LA. Diaphragm weakness in mechanically ventilated critically ill patients. Crit Care. 2013 Jun 20;17(3):R120. doi: 10.1186/cc12792. PMID 23786764
- [Background] Dres M, Dube BP, Mayaux J, Delemazure J, Reuter D, Brochard L, Similowski T, Demoule A. Coexistence and Impact of Limb Muscle and Diaphragm Weakness at Time of Liberation from Mechanical Ventilation in Medical Intensive Care Unit Patients. Am J Respir Crit Care Med. 2017 Jan 1;195(1):57-66. doi: 10.1164/rccm.201602-0367OC. PMID 27310484
- [Background] Zergeroglu MA, McKenzie MJ, Shanely RA, Van Gammeren D, DeRuisseau KC, Powers SK. Mechanical ventilation-induced oxidative stress in the diaphragm. J Appl Physiol (1985). 2003 Sep;95(3):1116-24. doi: 10.1152/japplphysiol.00824.2002. Epub 2003 May 30. PMID 12777408
- [Background] Maes K, Stamiris A, Thomas D, Cielen N, Smuder A, Powers SK, Leite FS, Hermans G, Decramer M, Hussain SN, Gayan-Ramirez G. Effects of controlled mechanical ventilation on sepsis-induced diaphragm dysfunction in rats. Crit Care Med. 2014 Dec;42(12):e772-82. doi: 10.1097/CCM.0000000000000685. PMID 25402297
- [Background] Powers SK, Hudson MB, Nelson WB, Talbert EE, Min K, Szeto HH, Kavazis AN, Smuder AJ. Mitochondria-targeted antioxidants protect against mechanical ventilation-induced diaphragm weakness. Crit Care Med. 2011 Jul;39(7):1749-59. doi: 10.1097/CCM.0b013e3182190b62. PMID 21460706
- [Background] Tang H, Shrager JB. The Signaling Network Resulting in Ventilator-induced Diaphragm Dysfunction. Am J Respir Cell Mol Biol. 2018 Oct;59(4):417-427. doi: 10.1165/rcmb.2018-0022TR. PMID 29768017
- [Background] Dridi H, Yehya M, Barsotti R, Reiken S, Angebault C, Jung B, Jaber S, Marks AR, Lacampagne A, Matecki S. Mitochondrial oxidative stress induces leaky ryanodine receptor during mechanical ventilation. Free Radic Biol Med. 2020 Jan;146:383-391. doi: 10.1016/j.freeradbiomed.2019.11.019. Epub 2019 Nov 19. PMID 31756525
- [Background] van den Berg M, Hooijman PE, Beishuizen A, de Waard MC, Paul MA, Hartemink KJ, van Hees HWH, Lawlor MW, Brocca L, Bottinelli R, Pellegrino MA, Stienen GJM, Heunks LMA, Wust RCI, Ottenheijm CAC. Diaphragm Atrophy and Weakness in the Absence of Mitochondrial Dysfunction in the Critically Ill. Am J Respir Crit Care Med. 2017 Dec 15;196(12):1544-1558. doi: 10.1164/rccm.201703-0501OC. PMID 28787181
- [Background] Aslan GK, Huseyinsinoglu BE, Oflazer P, Gurses N, Kiyan E. Inspiratory Muscle Training in Late-Onset Pompe Disease: The Effects on Pulmonary Function Tests, Quality of Life, and Sleep Quality. Lung. 2016 Aug;194(4):555-61. doi: 10.1007/s00408-016-9881-4. Epub 2016 Apr 22. PMID 27106274
- [Background] Vorona S, Sabatini U, Al-Maqbali S, Bertoni M, Dres M, Bissett B, Van Haren F, Martin AD, Urrea C, Brace D, Parotto M, Herridge MS, Adhikari NKJ, Fan E, Melo LT, Reid WD, Brochard LJ, Ferguson ND, Goligher EC. Inspiratory Muscle Rehabilitation in Critically Ill Adults. A Systematic Review and Meta-Analysis. Ann Am Thorac Soc. 2018 Jun;15(6):735-744. doi: 10.1513/AnnalsATS.201712-961OC. PMID 29584447
- [Background] Hearn E, Gosselink R, Freene N, Boden I, Green M, Bissett B. Inspiratory muscle training in intensive care unit patients: An international cross-sectional survey of physiotherapist practice. Aust Crit Care. 2022 Sep;35(5):527-534. doi: 10.1016/j.aucc.2021.08.002. Epub 2021 Sep 8. PMID 34507849
- [Background] Dres M, de Abreu MG, Merdji H, Muller-Redetzky H, Dellweg D, Randerath WJ, Mortaza S, Jung B, Bruells C, Moerer O, Scharffenberg M, Jaber S, Besset S, Bitter T, Geise A, Heine A, Malfertheiner MV, Kortgen A, Benzaquen J, Nelson T, Uhrig A, Moenig O, Meziani F, Demoule A, Similowski T; RESCUE-2 Study Group Investigators. Randomized Clinical Study of Temporary Transvenous Phrenic Nerve Stimulation in Difficult-to-Wean Patients. Am J Respir Crit Care Med. 2022 May 15;205(10):1169-1178. doi: 10.1164/rccm.202107-1709OC. PMID 35108175
- [Background] Dong Z, Liu Y, Gai Y, Meng P, Lin H, Zhao Y, Xing J. Early rehabilitation relieves diaphragm dysfunction induced by prolonged mechanical ventilation: a randomised control study. BMC Pulm Med. 2021 Mar 29;21(1):106. doi: 10.1186/s12890-021-01461-2. PMID 33781259
- [Background] Klompas M, Li L, Kleinman K, Szumita PM, Massaro AF. Associations Between Ventilator Bundle Components and Outcomes. JAMA Intern Med. 2016 Sep 1;176(9):1277-83. doi: 10.1001/jamainternmed.2016.2427. PMID 27428482
- [Background] Niel-Weise BS, Gastmeier P, Kola A, Vonberg RP, Wille JC, van den Broek PJ; Bed Head Elevation Study Group. An evidence-based recommendation on bed head elevation for mechanically ventilated patients. Crit Care. 2011;15(2):R111. doi: 10.1186/cc10135. Epub 2011 Apr 11. PMID 21481251
- [Background] Wang L, Li X, Yang Z, Tang X, Yuan Q, Deng L, Sun X. Semi-recumbent position versus supine position for the prevention of ventilator-associated pneumonia in adults requiring mechanical ventilation. Cochrane Database Syst Rev. 2016 Jan 8;2016(1):CD009946. doi: 10.1002/14651858.CD009946.pub2. PMID 26743945
- [Background] Pozuelo-Carrascosa DP, Cobo-Cuenca AI, Carmona-Torres JM, Laredo-Aguilera JA, Santacruz-Salas E, Fernandez-Rodriguez R. Body position for preventing ventilator-associated pneumonia for critically ill patients: a systematic review and network meta-analysis. J Intensive Care. 2022 Feb 22;10(1):9. doi: 10.1186/s40560-022-00600-z. PMID 35193688
- [Background] Spooner AJ, Corley A, Sharpe NA, Barnett AG, Caruana LR, Hammond NE, Fraser JF. Head-of-bed elevation improves end-expiratory lung volumes in mechanically ventilated subjects: a prospective observational study. Respir Care. 2014 Oct;59(10):1583-9. doi: 10.4187/respcare.02733. Epub 2014 May 20. PMID 24847096
- [Background] Brown C, Tseng SC, Mitchell K, Roddey T. Body Position Affects Ultrasonographic Measurement of Diaphragm Contractility. Cardiopulm Phys Ther J. 2018 Oct;29(4):166-172. doi: 10.1097/CPT.0000000000000083. Epub 2018 May 30. PMID 30319315
- [Background] Chang AT, Boots RJ, Hodges PW, Thomas PJ, Paratz JD. Standing with the assistance of a tilt table improves minute ventilation in chronic critically ill patients. Arch Phys Med Rehabil. 2004 Dec;85(12):1972-6. doi: 10.1016/j.apmr.2004.03.024. PMID 15605335
- [Background] Keogh C, Saavedra F, Dubo S, Aqueveque P, Ortega P, Gomez B, Germany E, Pinto D, Osorio R, Pastene F, Poulton A, Jarvis J, Andrews B, FitzGerald JJ. Non-invasive phrenic nerve stimulation to avoid ventilator-induced diaphragm dysfunction in critical care. Artif Organs. 2022 Oct;46(10):1988-1997. doi: 10.1111/aor.14244. Epub 2022 Apr 12. PMID 35377472
- [Background] Mezidi M, Guerin C. Effects of patient positioning on respiratory mechanics in mechanically ventilated ICU patients. Ann Transl Med. 2018 Oct;6(19):384. doi: 10.21037/atm.2018.05.50. PMID 30460258
- [Background] Hodgson CL, Stiller K, Needham DM, Tipping CJ, Harrold M, Baldwin CE, Bradley S, Berney S, Caruana LR, Elliott D, Green M, Haines K, Higgins AM, Kaukonen KM, Leditschke IA, Nickels MR, Paratz J, Patman S, Skinner EH, Young PJ, Zanni JM, Denehy L, Webb SA. Expert consensus and recommendations on safety criteria for active mobilization of mechanically ventilated critically ill adults. Crit Care. 2014 Dec 4;18(6):658. doi: 10.1186/s13054-014-0658-y. PMID 25475522
- [Background] Rosenfelder MJ, Helmschrott VC, Willacker L, Einhaupl B, Raiser TM, Bender A. Effect of robotic tilt table verticalization on recovery in patients with disorders of consciousness: a randomized controlled trial. J Neurol. 2023 Mar;270(3):1721-1734. doi: 10.1007/s00415-022-11508-x. Epub 2022 Dec 19. PMID 36536249
- [Background] Frazzitta G, Zivi I, Valsecchi R, Bonini S, Maffia S, Molatore K, Sebastianelli L, Zarucchi A, Matteri D, Ercoli G, Maestri R, Saltuari L. Effectiveness of a Very Early Stepping Verticalization Protocol in Severe Acquired Brain Injured Patients: A Randomized Pilot Study in ICU. PLoS One. 2016 Jul 22;11(7):e0158030. doi: 10.1371/journal.pone.0158030. eCollection 2016. PMID 27447483
- [Background] Yang X, Zhang T, Cao L, Ye L, Song W. Early Mobilization for Critically Ill Patients. Respir Care. 2023 Jun;68(6):781-795. doi: 10.4187/respcare.10481. Epub 2023 Apr 11. PMID 37041029